CLINICAL TRIAL: NCT05859646
Title: Evaluation of Streptococcus Mutans and Lactobacillus Species Due to Probiotic Use in Oral Flora
Brief Title: Effects of Probiotics on Streptococcus Mutans ve Lactobacillus Spp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Sakaryali Uyar (Other)
Responsible Party: Sponsor-Investigator, Didem Sakaryali Uyar, Asst. Prof. Dr., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-KA 19/41
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Tooth Decay; Probiotics; Streptococcus Mutans
Keywords: tooth caries; probiotics; qPCR; Streptococcus mutans; Lactobacillus
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: 2 separate groups, experimental and control, 6 month follow-up period, randomized distribution
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment was performed by a different researcher who was unaware of the group distributions in which patients were included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Group A-Probiotics group: Patients who started using probiotic drops after general anesthesia procedure
  Interventions: Dietary Supplement: Probiotic use
- Control (No Intervention): Group B-Control group: Patients who did not use any probiotics after general anesthesia procedure

INTERVENTIONS:
Dietary Supplement: Probiotic use — Probiotics were used for 3 months and all participated patients were followed for 6 months.
  Other Names: Follow-up after general anesthesia
  Arms: Probiotics

SUMMARY:
To evaluate the change of S. mutans and Lactobacillus spp. counts after all dental treatments were completed under general anesthesia and compare the groups in case of using probiotics and not using probiotics with the time for 6-months follow-up period.

DETAILED DESCRIPTION:
Fifthy-eight pediatric patients without any systemical diseases whose dental treatments were completed under general anesthesia were included in the study. The study was carried out as two-groups; Group A: Patients who started using probiotics after general anesthesia and Group B: Patients who did not use probiotics after general anesthesia. The counts of S. mutans and Lactobacillus spp. were determined by quantitative polymerase chain reaction (qPCR) by analysis of saliva samples taken from all patients on the day before the general anesthesia (T0), at 1-month (T1), 3-month (T2) and 6-month (T3) follow-up periods. The statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Every included child had at least 8 tooth with caries.

Exclusion Criteria:

* Patients who would not be able to give saliva samples due to high anxiety or lack of saliva were not included in this study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
S mutans count | 6 month
  CFU
Lactobacillus spp count | 6 month
  CFU

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is published, it can be sent to the individual upon reasonable request.

REFERENCES:
- [Derived] Sakaryali Uyar D, Uskudar Guclu A, Celik E, Memis Ozgul B, Altay Kocak A, Basustaoglu AC. Evaluation of probiotics' efficiency on cariogenic bacteria: randomized controlled clinical study. BMC Oral Health. 2024 Aug 2;24(1):886. doi: 10.1186/s12903-024-04659-y. PMID 39095860